CLINICAL TRIAL: NCT06940076
Title: Potential of Gayo Arabica Coffee Skin Extract Cream as a Topical Antioxidant: Clinical Trials on Humans
Brief Title: Potential of Gayo Arabica Coffee Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wahyu Lestari (Other)
Responsible Party: Sponsor-Investigator, Wahyu Lestari, Assistant Professor, Universitas Syiah Kuala
Organization: Universitas Syiah Kuala (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 094/ETIK-RSUDZA/2024
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- skin aging patients (Experimental)
  Interventions: Drug: gayo arabica coffee skin extract cream

INTERVENTIONS:
Drug: gayo arabica coffee skin extract cream — Assessment of glagou scale, skin analyzer, corneometer, and tewameter was done before and after the treatment . The subject will receive directions on how to use the cream before the study starts. The cream was used 2 times daily (7.40 AM and 1.00 PM) for 8 weeks.

SUMMARY:
The purpose of this study was to assess the effectiveness of gayo arabica coffee skin extract cream in the prevention of skin aging

ELIGIBILITY:
Inclusion Criteria:

* Women.
* have skin aging condition aged 30-60 years.
* Willing to participate in research based on research protocols.
* Before the research begins, research subjects are willing to sign informed consent and participate in the research until completion according to the research provisions from initial examination, re-control, and treatment until completion).

Exclusion Criteria:

* History of allergy to one of the ingredients in the cream.
* have a skin disorder and are undergoing treatment for skin disease.
* Undergoing treatment and use of facial cream in the last 1 month.
* History of allergy to coffee.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Glogau scale examination | 8 weeks from the beginning of the cream used by the subject
  the objective of this examination was to determine wrinkles. this parameter was measured before and after the study and then compared to assess the improvement
Skin analyzer examination | 8 weeks from the beginning of the cream used by the subject
  the objective of this examination was to determine skin moisture, pigmentation. this parameter was measured before and after the study and then compared to assess the improvement
Corneometer examination | 8 weeks from the beginning of the cream used by the subject
  the objective of this examination was to determine skin hydration. this parameter was measured before and after the study and then compared to assess the improvement

CONTACTS AND LOCATIONS:
Overall Officials: Wahyu Lestari, MD, Principal Investigator — Department of dermatology, venereology, and aesthetic dr. Zainoel Abidin General Hospital Banda Aceh, Nanggroe Aceh Darussalam, Indonesia
Locations (1):
- dr. Zainoel Abidin General Hospital, Banda Aceh, Special Region of Aceh, Indonesia

IPD SHARING:
Plan to Share IPD: No
to ensure the confidentiality of data obtained from respondents

REFERENCES:
- [Background] Esquivel P, Jiménez VM. Functional Properties of Coffee and Coffee By-products. Food Res Int. 2012;5(3):1-9. doi:10.1016/j.foodres.2011.05.028
- [Background] Murthy PS, Madhava Naidu M. Sustainable Management of Coffee Industry By-products and Value Addition - A review. Resour Conserv Recycl. Published online 2012:1-10. doi:10.1016/j.resconrec.2012.06.005
- [Background] Sholichah E, Apriani R, Desnilasari D, Karim MA. Produk Samping Kulit Kopi Arabika dan Robusta Sebagai Sumber Polifenol Untuk Antioksidan dan Antibakteri. Balai Besar Ind Has Perkeb. Published online 2019:57-66.
- [Background] Iriondo-DeHond A, Elizondo AS, Iriondo-DeHond M, Rios MB, Mufari R, Mendiola JA, Ibanez E, Castillo MDD. Assessment of Healthy and Harmful Maillard Reaction Products in a Novel Coffee Cascara Beverage: Melanoidins and Acrylamide. Foods. 2020 May 12;9(5):620. doi: 10.3390/foods9050620. PMID 32408584
- [Background] Ameca GM, Cerrilla MEO, Córdoba PZ, Cruz AD, Hernández MS, Haro JH. Chemical Composition and Antioxidant Capacity of Coffee Pulp. Cienc e Agrotecnologia. 2018;4(3):307-313. doi:10.1590/1413-70542018423000818
- [Background] Klingel T, Kremer JI, Gottstein V, Rajcic de Rezende T, Schwarz S, Lachenmeier DW. A Review of Coffee By-Products Including Leaf, Flower, Cherry, Husk, Silver Skin, and Spent Grounds as Novel Foods within the European Union. Foods. 2020 May 21;9(5):665. doi: 10.3390/foods9050665. PMID 32455549
- [Background] Tuong W, Walker L, Sivamani RK. Polyphenols as novel treatment options for dermatological diseases: A systematic review of clinical trials. J Dermatolog Treat. 2015;26(4):381-8. doi: 10.3109/09546634.2014.991675. Epub 2014 Dec 30. PMID 25424055
- [Background] Islam MT, Tabrez S, Jabir NR, Ali M, Kamal MA, da Silva Araujo L, De Oliveira Santos JV, Da Mata AMOF, De Aguiar RPS, de Carvalho Melo Cavalcante AA. An Insight into the Therapeutic Potential of Major Coffee Components. Curr Drug Metab. 2018;19(6):544-556. doi: 10.2174/1389200219666180302154551. PMID 29512445
- [Background] Petruk G, Del Giudice R, Rigano MM, Monti DM. Antioxidants from Plants Protect against Skin Photoaging. Oxid Med Cell Longev. 2018 Aug 2;2018:1454936. doi: 10.1155/2018/1454936. eCollection 2018. PMID 30174780
- [Background] Bosch R, Philips N, Suarez-Perez JA, Juarranz A, Devmurari A, Chalensouk-Khaosaat J, Gonzalez S. Mechanisms of Photoaging and Cutaneous Photocarcinogenesis, and Photoprotective Strategies with Phytochemicals. Antioxidants (Basel). 2015 Mar 26;4(2):248-68. doi: 10.3390/antiox4020248. PMID 26783703